CLINICAL TRIAL: NCT00769782
Title: Phase II Multicenter Clinical Trial on Surgery for Patients With Resectable Hepatic Metastasis From Gastrointestinal Stromal Tumors (GISTs)
Brief Title: Surgery in Treating Patients With Liver Metastasis From a Gastrointestinal Stromal Tumor
Acronym: GISTs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Niigata University Medical & Dental Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000615624; NIIGATAU-TRIGIST0804 (Other: Niigata University Medical and Dental Hospital)
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Gastrointestinal Stromal Tumor; Metastatic Cancer
Keywords: gastrointestinal stromal tumor; liver metastases
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- therapeutic conventional surgery (Experimental): All patients undergo suegery to achieve macroscopic complete resection within 28 days after enrollment (including enrollment day). As long as tumor free margin is ensured, all resection margin distances and all surgical procedure are accepted. Surgical treatment in this study excludes the following, radiofrequency ablation (RFA) without resection of liver only or microwave coagulation therapy (MCT) only; for RFA or MCT is used as additional treatment under judgment of primary physician for new liver tumor which comfirmed during surgery in different parts of liver except portion scheduled for resection, RFA and MCT are included. After histological curative resection, patients are observed without treatment until comfirming recurrence. Patients with incomplete tumor removal are withdrawn from protcol treatment and receive imatinib treatment, 400 mg/day orally. For reccurrence is comfirmed, patients receive imatinib treatment, 400 mg/day orally.
  Interventions: Procedure: therapeutic conventional surgery

INTERVENTIONS:
Procedure: therapeutic conventional surgery — All patients undergo suegery to achieve macroscopic complete resection within 28 days after enrollment (including enrollment day). As long as tumor free margin is ensured, all resection margin distances and all surgical procedure are accepted. Surgical treatment in this study excludes the following, radiofrequency ablation (RFA) without resection of liver only or microwave coagulation therapy (MCT) only; for RFA or MCT is used as additional treatment under judgment of primary physician for new liver tumor which comfirmed during surgery in different parts of liver except portion scheduled for resection, RFA and MCT are included. After histological curative resection, patients are observed without treatment until comfirming recurrence. Patients with incomplete tumor removal are withdrawn from protcol treatment and receive imatinib treatment, 400 mg/day orally. For reccurrence is comfirmed, patients receive imatinib treatment, 400 mg/day orally.

SUMMARY:
RATIONALE: Surgery may be an effective treatment for liver metastasis from a gastrointestinal stromal tumor.

PURPOSE: This phase II trial is studying how well surgery works in treating patients with liver metastasis from a gastrointestinal stromal tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the safety and efficacy of surgery in patients with resectable hepatic metastasis secondary to gastrointestinal stromal tumor.

OUTLINE: This is a multicenter study.

Patients undergo surgical resection of hepatic metastasis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of gastrointestinal stromal tumor (GIST)
* Hepatic metastasis meeting the following criteria:

  * Clinically diagnosed as surgically resectable with no macroscopic residual tumor
  * No more than 3 hepatic metastases
  * Synchronous hepatic metastasis allowed provided primary tumor is also resectable
  * Does not require radiofrequency ablation and/or microwave coagulation therapy to control the disease
* No extrahepatic metastasis
* No history of GIST recurrence

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Leukocyte count ≥ 3,000/μL
* Neutrophil count ≥ 1,500/μL
* Hemoglobin ≥ 8.0 g/dL
* Platelet count ≥ 75,000/μL
* Total bilirubin ≤ 2.0 mg/dL
* ALT and AST < 120 IU/L
* GTP < 210 IU/L
* Not pregnant
* No poorly controlled diabetes mellitus
* No NYHA class III-IV cardiac function
* No hepatitis B or hepatitis B carriers
* No other malignancy requiring treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior interventional radiology for metastatic disease
* No prior or concurrent imatinib mesylate
* No other concurrent treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival | 7.5 years
  Recurrence-free survival is defined as time from date of surgery until date of recurrence or death from any cause, whichever comes first.

SECONDARY OUTCOMES:
Overall survival | 7.5 years
  Overall survival is defined as time from date of surgery until date of death from any cause.
Histological curative resection | At surgery
  Histological curative resection is defined as complete tumor removal which comfirmed by pathological assessment of resected tissue. For radiofrequency ablation (RFA) or microwave coagulation therapy (MCT) is used as additional treatment for the new liver tumor which confirmed during surgery in different parts of liver except the portion scheduled for resection, the case is regarded as incomplete resection (R1). For peritoneal metastasis is confirmed during surgery, the case is regarded as incomplete resection (R1) regardless of macroscopic complete resection.
Types and severities of adverse events | 7.5 years
  Types and severities of adverse events from date of starting protocol treatment until 30 days after date of finishing the treatment are evaluated according to Japanese version of the National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0) by Translational Research Informatics Center.

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuo Kanda, MD, Principal Investigator — Niigata University Medical & Dental Hospital
Locations (37):
- Japan (37):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - Aichi Medical University, Nagoya, Aichi-ken
  - Hirosaki University, School of Medicine, Hirosaki, Aomori
  - National Hospital Organization Kure Medical Center, Kure, Hiroshima
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Iwate Medical University Hospital, Morioka, Iwate
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - International Goodwill Hospital, Yokohama, Kanagawa
  - Kochi Medical School, Nankoku, Kochi
  - Kyoto Second Red Cross Hospital, Kanigyou-ku, Kyoto
  - University of Miyazaki Hospital, Kiyotake, Miyazaki
  - Niigata Prefectural Central Hospital, Jōetsu, Niigata
  - Nagaoka Chuo General Hospital, Nagaoka, Niigata
  - Kawasaki Medical School, Kurashiki, Okayama-ken
  - Ryukyu University Hospital, Nishiharacho, Okinawa
  - Sakai Municipal Hospital, Sakai, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Toyonaka Municipal Hospital, Toyonaka, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Hamamatsu University School of Medicine, Hamamatsu, Shizuoka
  - University of Yamanashi Hospital, Chūō, Yamanashi
  - Kyushu University Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Kagoshima University, Kagoshima
  - Kimitsu Chuo Hospital, Kisarazu
  - Kochi Health Sciences Center, Kochi
  - Kumamoto University Hospital, Kumamoto
  - Niigata University Medical and Dental Hospital, Niigata
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Juntendo University Shizuoka Hospital, Shizuoka
  - Shizuoka Cancer Center, Shizuoka
  - Tokushima University Hospital, Tokushima
  - Tokyo Metropolitan - Komagome Hospital, Tokyo
  - Keio University Hospital, Tokyo
  - Toyama University Hospital, Toyama
  - Yamagata University Hospital, Yamagata